CLINICAL TRIAL: NCT00760240
Title: Objective Evaluation of the Ability of Patients With Decreased Vision or Restricted Visual Fields to Properly Instill Eye Drops
Brief Title: Ability of Patients With Low Vision to Properly Instill Eye Drops
Status: Completed | Type: Observational
Sponsor: Mid-Atlantic Glaucoma Experts (Other)
Responsible Party: Amy L Hennessy, Mid-Atlantic Glaucoma Experts
Other Study IDs: SI-08-64
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Glaucoma; Retinal Pathology
Keywords: compliance; eyedrop instillation; How patients with low vision due to glaucoma or retinal pathology instill eyedrops into their own eyes.
MeSH Terms: conditions — Glaucoma; Patient Compliance

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glaucoma patients: This is a group of patients with restricted visual fields or ETDRS visual acuity of 20/60 or worse
- Retina patients: A group of patients with retinal pathology(ARMD, CME, diabetic retinopathy) contributing to their decreased vision.

SUMMARY:
The investigators are interested in seeing how people with low vision (decreased visual acuity or restricted visual fields) instill eye drops into their own eyes. The investigators hypothesis is that this population will have more difficulty with self-instillation of drops than a better-seeing population. The investigators aim to explore whatever factors may be involved in preventing this population from getting prescribed eyedrops into their eyes, whether it is more related to visual field or visual acuity.

DETAILED DESCRIPTION:
This is a study that involves a questionnaire that a study participant fills out, detailing their experience with eyedrops (if any), followed by a video recording of them instilling artificial tears into their worse-seeing eye, with their dominant hand. Patients must have visual acuity worse than 20/60 in at least one eye, and/or have a recent visual field that demonstrated Hodapp criteria for Moderate or Severe visual field damage. This is an observational study of how patients with low vision due to either glaucoma or retinal disease instill eyedrops. Each video will be "graded" by the principal investigator for "success" at instilling eyedrops, and patients will be stratified by their visual acuity or visual field, and whether they have a primary diagnosis of glaucoma or retinal disease.

ELIGIBILITY:
Inclusion Criteria:

* ETDRS visual acuity 20/60 or worse

Exclusion Criteria:

* Unwilling to participate
* Light perception vision
* No light perception vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients reporting for appointments at outpatients referral practices shared by 2 glaucoma and 3 retina specialists
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Successful instillation of a single eyedrop onto the surface of the eye | 2 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Glaucoma Specialists/Retina Care Center, Baltimore, Maryland, United States